CLINICAL TRIAL: NCT01247714
Title: Clinical Evaluation of a Specific Enteral Diet for Diabetics.A Randomised Cross-Over Study
Brief Title: Clinical Evaluation of a Specific Enteral Diet for Diabetics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vegenat, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: VEGENAT-DIABET NP UGR; DIABET NP 2009-PROYECTO CDTI (Other: VEGENAT, S.A.)
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2010-11

CONDITIONS: Hyperglycemia; Diabetics; Metabolic Syndrome
Keywords: T-Diet plus Diabet NP; Diabetic; Enteral Nutrition; Glycaemic response; Metabolic Syndrome; Insulin resistance; Lipidic profile
MeSH Terms: conditions — Hyperglycemia; Metabolic Syndrome; Insulin Resistance | interventions — Phentermine; Glucerna

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): The group 1 will receive the experimental product T-Diet plus Diabet NP for the first month followed by a reference diet corresponding to a current marketed product (Glucerna SR, Abbott) for the second month, then the patients will receive a control product non specific for diabetic patients (T-Diet plus Standard)for the third month, and finally a specific diet for diabetic patients (Novasource, Nestlé Healthcare Nutrition)for the fourth month.
  Interventions: Dietary Supplement: T-Diet plus Standard; Dietary Supplement: T-Diet plus Diabet NP; Dietary Supplement: Glucerna; Dietary Supplement: Novasource
- Group 2 (Active Comparator): The group 2 will receive a reference diet corresponding to a current marketed product (Glucerna SR, Abbott)for the first month, followed by the experimental product T-Diet plus Diabet NP for the second month, then the patients will receive a specific diet for diabetic patients (Novasource, Nestlé Healthcare Nutrition)for the third month, and finally a control product non specific for diabetic patients (T-Diet plus Standard)for the fourth month
  Interventions: Dietary Supplement: T-Diet plus Standard; Dietary Supplement: T-Diet plus Diabet NP; Dietary Supplement: Glucerna; Dietary Supplement: Novasource

INTERVENTIONS:
Dietary Supplement: T-Diet plus Standard — T-Diet plus Standard is a complete balanced protein and energy oral nutrition supplement, indicated for the dietary management of patients with related malnutrition.
  Other Names: PLUS STD
Dietary Supplement: T-Diet plus Diabet NP — T-Diet plus Diabet NP is a complete balanced oral nutrition supplement, indicated for the dietary management of diabetic patients or hyperglycemia related malnutrition.
  Other Names: DIABET NP
Dietary Supplement: Glucerna — GLUCERNA 1.0 CAL is a reduced-carbohydrate, modified-fat, fiber-containing formula clinically shown to blunt blood-glucose response in patients with abnormal glucose tolerance.
  Other Names: GLCR
Dietary Supplement: Novasource — Complete high protein diet for diabetic patients and hyperglycemic
  Other Names: NVS

SUMMARY:
The hypothesis of the proposed trials is that the regular intake of a specific diet designed for enteral nutrition of type 2 diabetic patients results into a better nutritional status. Thus, the aim of the study is to scientifically evaluate the healthy effects of the administration of an enteral complete diet for diabetic patients (T-Diet plus Diabet).

DETAILED DESCRIPTION:
This new complete diet has been carefully formulated, and incorporates functional ingredients based on:

1. A good gastrointestinal and metabolic tolerance of the product.
2. Beneficial outcomes in the nutritional status.
3. A good control of the glycaemic response and the lipidic profile, allowing an improvement of metabolic syndrome and insulin resistance indicators and hunger-satiety regulation.

The experimental enteral product is a complete diet that includes, as carbohydrates, high-molecular maltodextrin, resistant maltodextrin, fructooligosaccharides and cellulose, and does not contain added fructose. Indeed, this product contains eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA).

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Subjects older than 55 years.
* Male or female
* Requirement of total enteral nutrition (TEN) during at least 3 months.
* Under medical supervision.
* Voluntary informed consent for participation.

Exclusion Criteria:

* Unstable clinical situation
* Fatal illness
* Patients treated with lipidic drugs
* Refusal to participate in the study or being enrolled in other clinical trials.
* Social or humanitarian reason

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Nutritional status and Glycaemia | 9 months
  * Evaluation of the nutritional status of diabetic patients fed the T-Diet Plus Diabet NP in comparison with the reference and the control diet.
  * Evaluation of glycaemia and glycosylated hemoglobin

SECONDARY OUTCOMES:
Biochemicals parameters measure | 9 months
  * Confirmation of gastrointestinal tolerance of the product
  * To assess changes in glycaemic response and lipidic profile in theses patients in relation with the diet, including parameters characteristic of metabolic syndrome, insulin resistace and hunger-satiety mechanism.
  * To analyse changes of incretins and gastrointestinal peptides levels.
  * To compare inflammatory and endothelial damage markers related with cardiovascular morbidity.
  * Genotyping and gene expression analysis of genes related with diabetes and insulin resistance

CONTACTS AND LOCATIONS:
Overall Officials: Ángel Gil, PhD, Principal Investigator — Departament of Biochemistry and Molecular Biology II. University of Granada
Locations (1):
- Department of Biochemistry and Molecular Biology II. University of Granada, Granada, Granada, Spain